CLINICAL TRIAL: NCT04417465
Title: A Phase 1, Multi-center, Open Label First-in-Human Study With ABBV-CLS-579 Alone and in Combination in Subjects With Locally Advanced or Metastatic Tumors
Brief Title: First In Human Study With ABBV-CLS-579 When Given Alone and In Combination In Participants With Locally Advanced Or Metastatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-124; 2020-000639-28 (EudraCT Number)
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Cancer; Tumor; ABBV-CLS-579; PD-1; VEGFR TKI; ccRCC; NSCLC; MSI-H; HNSCC
MeSH Terms: conditions — Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Monotherapy Dose Escalation (Experimental): ABBV-CLS-579 will be administered as a monotherapy in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-579
- Combination Dose Escalation with PD-1 (Experimental): ABBV-CLS-579 will be administered in combination with Programmed Cell Death-1 Inhibitor in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-579; Drug: PD-1 inhibitor
- Backfill Cohorts with Monotherapy (Experimental): ABBV-CLS-579 will be administered as a monotherapy in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-579
- Backfill Cohorts in Combination with PD-1 (Experimental): ABBV-CLS-579 will be administered in combination with Programmed Cell Death-1 Inhibitor in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-579; Drug: PD-1 inhibitor
- Combination Expansion with PD-1 (Experimental): ABBV-CLS-579 will be administered at the determined recommended dose in subjects with locally advanced or metastatic, relapsed or refractory head and neck squamous cell carcinoma (HNSCC), relapsed or refractory non-small cell lung cancer (NSCLC), microsatellite instability-high (MSI-H) tumors, and advanced clear cell renal cell carcinoma (ccRCC)
  Interventions: Drug: ABBV-CLS-579; Drug: PD-1 inhibitor
- Combination Expansion with VEGFR TKI (Experimental): ABBV-CLS-579 will be administered at the determined recommended dose in combination with Vascular Endothelial Growth (VEGFR) Factor Receptor Tyrosine Kinase Inhibitor (TKI) in subjects with advanced ccRCC.
  Interventions: Drug: ABBV-CLS-579; Drug: VEGFR TKI

INTERVENTIONS:
Drug: ABBV-CLS-579 — Oral Capsule
Drug: PD-1 inhibitor — Intravenous (IV) infusion
  Arms: Backfill Cohorts in Combination with PD-1; Combination Dose Escalation with PD-1; Combination Expansion with PD-1
Drug: VEGFR TKI — Oral Tablet
  Arms: Combination Expansion with VEGFR TKI

SUMMARY:
The purpose of this study is to see how safe and effective ABBV-CLS-579 is when used alone and in combination with a PD-1 target agent or with a VEGF TKI.

ABBV-CLS-579 is an investigational drug being developed for the treatment of tumors.

The trial aims to establish a safe, tolerable, and efficacious dose of ABBV-CLS-579 as monotherapy and in combination. The study will be conducted in three parts. Part 1 Monotherapy Dose Escalation, Part 2 Combination Dose Escalation, and Part 3 Combination Dose Expansion.

Part 1, ABBV-CLS-579 will be administered alone in escalating dose levels to eligible subjects who have advanced solid tumors.

Part 2, ABBV-CLS-579 will be administered at escalating dose levels in combination with a PD-1 targeting agent to eligible subjects who have advanced solid tumors.

Part 3, ABBV-CLS-579 will be administered at the determined recommended dose in combination with a PD-1 target agent or with a VEGFR TKI in subjects with locally advanced or metastatic, relapsed or refractory head and neck squamous cell carcinoma (HNSCC), relapsed or refractory non-small cell lung cancer (NSCLC), and advanced clear cell renal cell carcinoma (ccRCC).

Adult participants with a diagnosis of some solid tumors for which no effective standard therapy exists or has failed will be enrolled. Participants will receive study treatment until disease progresses or discontinued.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must weigh at least 35 kilograms (kg).
* For Monotherapy and Combination Dose Escalation:

  * Histologically or cytologically proven metastatic or locally advanced tumors (with measurable disease defined by Response Evaluation Criteria In Solid Tumors [RECIST] v1.1), for which no effective standard therapy exists, or where standard therapy has failed. Participants must have received at least 1 prior systemic anticancer therapy for the indication being considered.
* For Combination Dose Expansion:

  * For the following tumor types, the subject must have received at least 1 prior line containing PD-1/PD-L1 target therapy.

Indication with outcome of Prior PD-1/PD-L1 Targeted Therapy and other disease characteristics:

* NSCLC

  * Relapsed: Tumors express PD-L1 (TPS ≥ 1%) as determined by the FDA-approved Agilent PD-L1 IHC 22C3 pharmDx kit
  * Refractory: Tumors express PD-L1 (TPS ≥ 1%) as determined by the FDA-approved Agilent PD-L1 IHC 22C3 pharmDx kit
* ccRCC

  * Relapsed or Refractory: Advanced disease (locally advanced or metastatic)
* MSI-H tumors

  * Refractory: Locally advanced or metastatic MSI-H tumors whose tumors are determined to have a MSI-H status by PCR or NGS tests, or dMMR by IHC tests.
* HNSCC

  * Relapsed or Refractory: Tumors express PD-L1 (CPS ≥ 1] as determined by the FDA approved PD-L1 Agilent IHC 22C3 pharmDx kit
* For Combination Dose Expansion:

  * Locally advanced or metastatic, advanced ccRCC who have relapsed after at least 1 prior VEGFR TKI therapy
* Received at least 1 prior line containing PD 1/PD L1 targeted therapy with a best response by RECIST v1.1 of CR/PR (any duration) or stable disease (for greater than 6 months)
* Received at least 1 prior line containing PD-1/PD-L1 targeted therapy and have had disease progression (in the absence of best response of CR/PR/stable disease by RECIST v1.1) with PD 1/PD L1 targeted therapy
* An Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Life expectancy of ≥ 12 weeks.
* Laboratory values meeting protocol criteria.
* If the subject is on anticoagulant therapy, INR must be within therapeutic goal.
* QT interval corrected for heart rate < 450 msec (using Fridericia's correction), and no clinically significant electrocardiographic findings.

Exclusion Criteria:

* Untreated brain or meningeal metastases (participants with history of metastases are eligible provide they do not require ongoing steroid treatment and have shown clinical and radiographic stability for at least 28 days after definitive therapy).
* Unresolved Grade 2 or higher toxicities related to previous anticancer therapy except alopecia.
* History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
* Recent history (within 6 months) of congestive heart failure (defined as New York Heart Association, Class 2 or higher), ischemic cardiovascular event, pericarditis, or clinically significant pericardial effusion, cardiac arrythmia or peripheral artery disease.
* Recent history (within 6 months) of Childs-Pugh B or C classification of liver disease.
* History of clinically significant medical and/or psychiatric conditions or any other reason that, in the opinion of the investigator, would interfere with participation in this study or would make the participant an unsuitable candidate to receive study drug.
* History of uncontrolled, clinically significant endocrinopathy.
* Known gastrointestinal disorders making absorption of oral medications problematic. Inability to swallow capsules.
* If treated with anti-programmed cell death protein-1 (aPD-1)/antiprogrammed cell death protein-ligand 1(aPD-L1) targeting or other immunostimulatory agents in the past: excluded if had prior pneumonitis, prior Grade 3 or higher immune mediated toxicity, hypersensitivity to administered drug or drug related toxicity requiring discontinuation.
* Active autoimmune disease requiring systemic treatment in past 2-years (exceptions for endocrinopathies, vitiligo or atopic conditions)
* History of solid organ transplant or allogeneic stem cell transplant.
* History of interstitial lung disease or pneumonitis.
* Major surgery ≤ 28 days prior to first dose of study drug.
* Poorly controlled hypertension
* History of hemorrhage, including hemoptysis, hematemesis, or melena
* History of other malignancy, with the following exceptions:

  * No known active disease present for within 3 years before first dose of study treatment and felt to be at low recurrence by investigator
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection per local testing practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma/Serum Concentration (Cmax) Of ABBV-CLS-579 | Baseline Up to Approximately Day 44
  Maximum plasma/serum concentration of ABBV-CLS-579
Maximum Observed Plasma/Serum Concentration (Cmax) Of Metabolite M4 | Baseline Up to Approximately Day 44
  Maximum plasma/serum concentration of Metabolite M4
Maximum Observed Plasma/Serum Concentration (Cmax) Of PD-1 Inhibitor | Baseline Up to Approximately Day 64
  Maximum plasma/serum concentration of PD-1 inhibitor
Maximum Observed Plasma/Serum Concentration (Cmax) Of VEGFR TKI | Baseline Up to Approximately Day 64
  Maximum plasma/serum concentration of VEGFR TKI
Time To Cmax (Tmax) Of ABBV-CLS-579 | Baseline Up to Approximately Day 44
  The amount of time taken to reach Cmax
Time To Cmax (Tmax) Of Metabolite M4 | Baseline Up to Approximately Day 44
  The amount of time taken to reach Cmax
Time To Cmax (Tmax) Of PD-1 Inhibitor | Baseline Up to Approximately Day 64
  The amount of time taken to reach Cmax
Time To Cmax (Tmax) Of VEGFR TKI | Baseline Up to Approximately Day 64
  The amount of time taken to reach Cmax
Terminal Phase Elimination Rate Constant (β) Of ABBV-CLS-579 | Baseline Up to Approximately Day 44
  Terminal phase elimination rate constant (β or Beta)
Terminal Phase Elimination Rate Constant (β) Of Metabolite M4 | Baseline Up to Approximately Day 44
  Terminal phase elimination rate constant (β or Beta)
Terminal Phase Elimination Rate Constant (β) Of PD-1 Inhibitor | Baseline Up to Approximately Day 64
  Terminal phase elimination rate constant (β or Beta)
Terminal Phase Elimination Rate Constant (β) Of VEGFR TKI | Baseline Up to Approximately Day 64
  Terminal phase elimination rate constant (β or Beta)
Terminal Phase Elimination Half-Life (t1/2) Of ABBV-CLS-579 | Baseline Up to Approximately Day 44
  Terminal phase elimination half-life (t1/2)
Terminal Phase Elimination Half-Life (t1/2) Of Metabolite M4 | Baseline Up to Approximately Day 44
  Terminal phase elimination half-life (t1/2)
Terminal Phase Elimination Half-Life (t1/2) Of PD-1 Inhibitor | Baseline Up to Approximately Day 64
  Terminal phase elimination half-life (t1/2)
Terminal Phase Elimination Half-Life (t1/2) Of VEGFR TKI | Baseline Up to Approximately Day 64
  Terminal phase elimination half-life (t1/2)
Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of ABBV-CLS-579 | Baseline Up to Approximately Day 44
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of Metabolite M4 | Baseline Up to Approximately Day 44
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of PD-1 Inhibitor | Baseline Up to Approximately Day 64
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of VEGFR TKI | Baseline Up to Approximately Day 64
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Recommended Expansion Dose and/or Maximum Tolerated Dose of ABBV-CLS-579 | Baseline through Study Completion (approximately 3 years)
  The Expansion Dose and/or MTD of ABBV-CLS-579 will be determined during the monotherapy dose escalation phase of the study
Recommended Expansion Dose and/or Maximum Tolerated Dose of ABBV-CLS-579 and a PD-1 Inhibitor | Baseline through Study Completion (approximately 3 years)
  The Expansion Dose and/or MTD of ABBV-CLS-579 and PD-1 inhibitor will be determined during the combination therapy dose escalation phase of the study
Objective Response Rate (ORR) Of ABBV-CLS-579 And PD-1 Targeting Agent Base On Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, of ABBV-CLS-579 in locally or metastatic HNSCC, NSCLC, MSI-H tumors, and advanced ccRCC | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Objective Response Rate (ORR) on RECIST v1.1, of ABBV-CLS-579 administered in combination with VEGFR TKI in advanced ccRCC | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Of ABBV-CLS-579 And PD-1 Targeting Agent Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Objective Response Rate (ORR) Of ABBV-CLS-579 Monotherapy Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Best Overall Response (BOR) Of ABBV-CLS-579 Monotherapy Based On RECIST v1.1 | Baseline through Study Completion (approximately 3 years)
  BOR is defined as the best response recorded from the start of the treatment until disease progression/recurrence
Best Overall Response (BOR) Of ABBV-CLS-579 And PD-1 Targeting Agent Based On RECIST v1.1 | Baseline through Study Completion (approximately 3 years)
  BOR is defined as the best response recorded from the start of the treatment until disease progression/recurrence
Change from Baseline QTc | Baseline through Study Completion (approximately 3 years)
  QT prolongation is measured by the QT interval measurement corrected for heart rate (QTc) change from baseline

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - Highlands Oncology Group Springdale, Springdale, Arkansas
  - Yale University, New Haven, Connecticut
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
- France (2):
  - Hopital Saint-Andre, Bordeaux
  - Institut Gustave Roussy, Villejuif
- The Chaim Sheba Medical Center, Ramat Gan, Israel
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-Shi, Chiba
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Seoul National University Hospital, Seoul, South Korea
- Spain (4):
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No